CLINICAL TRIAL: NCT07085910
Title: Modulating Interhemispheric Interactions Using Hebbian-Type Associative Stimulation to Promote Upper Extremity Motor Recovery Following Stroke
Brief Title: Hebbian-Type Associative Stimulation in Stroke Rehabilitation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSEARS20240927001
Record Dates: First submitted 2025-07-17; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-06

CONDITIONS: Stroke
Keywords: Stroke; Neuromodulation; Transcranial magnetic stimulation; Upper extremity; Rehabilitation and Occupational Therapy
MeSH Terms: conditions — Stroke | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Corticocortical paired associative stimulation (ccPAS) (Experimental): The ccPAS will be applied using two MagPro X100 stimulators connected to two vertically oriented figure-of-eight coils designed for bilateral hemispheric stimulation. Each ccPAS session will involve the delivery of 90 paired pulses, stimulating the M1s over both the contralesional and ipsilesional hemispheres at a frequency of 0.05 Hz. Each session will be 30 minutes, and the interstimulus interval between paired pulses will be 8 ms to ensure that the ipsilesional M1 neurons are always activated before the firing of contralesional M1 neurons.
  Interventions: Device: Transcranial magnetic stimulation - dual coil
- Conventional single-site low frequency repetitive transcranial magnetic stimulation (rTMS) (Active Comparator): LF rTMS will be performed using a TMS stimulator and the same stimulation coil (MC-B65-HO). The stimulation target will be set the contralesional M1 area, determined using motor hotspot hunting. In line with our recent trial, a total of 1200 pulses (20 mins) with a frequency of 1 Hz and an intensity of 120% of the RMT will be delivered to the contralesional M1
  Interventions: Device: Transcranial magnetic stimulation
- Sham corticocortical paired associative stimulation (ccPAS) (Sham Comparator): The same dual-coil setup (MC-B65-HO) and stimulation intensity during sham stimulation as in the ccPAS group will be utilized. However, the inter-stimulus interval between paired pulses will be adjusted to 100 ms (a duration that prevents any STDP-like effects from being induced by repetitive paired-pulse stimulation)
  Interventions: Device: Transcranial magnetic stimulation - dual coil

INTERVENTIONS:
Device: Transcranial magnetic stimulation - dual coil — The dual coil stimulation will be applied using two MagPro X100 stimulators connected to two vertically oriented figure-of-eight coils designed for bilateral hemispheric stimulation.
  Arms: Corticocortical paired associative stimulation (ccPAS); Sham corticocortical paired associative stimulation (ccPAS)
Device: Transcranial magnetic stimulation — Single coil TMS will be performed using a TMS stimulator and the same stimulation coil (MC-B65-HO).
  Arms: Conventional single-site low frequency repetitive transcranial magnetic stimulation (rTMS)

SUMMARY:
Stroke remains the primary cause of long-term neurological disabilities. Effective rehabilitation solutions are essential to alleviate the burden poststroke survivors impose on hospitals and community services. Following unilateral stroke, interhemispheric balance is disrupted. Prior studies have extensively documented that exaggerated interhemispheric inhibitory flow from the contralesional to the ipsilesional hemisphere prevents maximal functional recovery in poststroke survivors. Therefore, we aimed to test the modulatory effects of a Hebbian-type plasticity induction paradigm using corticocortical paired associative stimulation (ccPAS) over the bilateral motor cortex. This approach aims to reverse the abnormal inhibitory flow from the contralesional to the ipsilesional hemisphere and assess its clinical benefits on upper extremity motor recovery in patients with stroke. In this randomized controlled trial, we hypothesize that Hebbian-type ccPAS would be more effective than sham ccPAS and conventional single-site inhibitory rTMS delivered to the contralesional hemisphere at improving hemiplegic upper limb motor functionality and modulating interhemispheric activity to an equilibrium state among patients with stroke. This approach seeks to address diseases related to brain network impairments, such as stroke. This project will provide insights into the recovery mechanisms activated following neurological diseases from the perspective of the Hebbian learning rules of associative plasticity.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis with monohemispheric ischemic subcortical stroke (with intact corpus callosum), with stroke onset ≥6 months,
2. Age 40-75 years.
3. Residual upper limb function between levels 3-6, according to the Functional Test for the Hemiplegic Upper Extremity (FTHUE), indicating mildly to moderately impaired upper limb motor function.
4. Capable of providing informed written consent.

Exclusion Criteria:

1. any contraindications for TMS (screened using the safety checklist by Rossi)
2. Diagnosis of any concomitant neurological diseases other than stroke.
3. Signs of cognitive impairment, defined as a Montreal cognitive assessment Hong Kong version score <21/22 out of 30 .
4. Severe spasticity in the hemiparetic upper limb muscles, with a Modified Ashworth score >2.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-07-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
The Fugl-Meyer Assessment-Upper Extremity Scores | Baseline
  The Fugl-Meyer Assessment-Upper Extremity Scores (FMA-UE) is the gold standard for assessing poststroke upper limb motor control. It is used to determine the movement, coordination, and reflex action of the affected upper limb in poststroke people.
The Fugl-Meyer Assessment-Upper Extremity Scores | At 4 weeks
  The Fugl-Meyer Assessment-Upper Extremity Scores (FMA-UE) is the gold standard for assessing poststroke upper limb motor control. It is used to determine the movement, coordination, and reflex action of the affected upper limb in poststroke people.
The Fugl-Meyer Assessment-Upper Extremity Scores | At 3-month
  The Fugl-Meyer Assessment-Upper Extremity Scores (FMA-UE) is the gold standard for assessing poststroke upper limb motor control. It is used to determine the movement, coordination, and reflex action of the affected upper limb in poststroke people.

SECONDARY OUTCOMES:
Interhemispheric signal propagation (ISP) in TMS-evoked potential | Baseline
  ISP measured using concurrent TMS-evoked potential is set as another outcome for measuring the interhemispheric inhibitory flow between the bilateral M1s. TMS-evoked activity will be defined as the local mean field power (LMFP) of six channels surrounding the M1 (Left: C1, C3, C5, CP1, CP3, CP5; Right: C2, C4, C6, CP2, CP4, CP6) in a specific time frame. Because of the approximately 10 ms of transcallosal conduction, the LMFP from 50 to 130 ms is rectified for the stimulated M1 and from 60 to 140 ms for the non-stimulated M1. A higher ISP value indicates a higher inhibitory flow from the non-stimulated M1 to the stimulated M1.
Interhemispheric signal propagation (ISP) in TMS-evoked potential | At 4-week
  ISP measured using concurrent TMS-evoked potential is set as another outcome for measuring the interhemispheric inhibitory flow between the bilateral M1s. TMS-evoked activity will be defined as the local mean field power (LMFP) of six channels surrounding the M1 (Left: C1, C3, C5, CP1, CP3, CP5; Right: C2, C4, C6, CP2, CP4, CP6) in a specific time frame. Because of the approximately 10 ms of transcallosal conduction, the LMFP from 50 to 130 ms is rectified for the stimulated M1 and from 60 to 140 ms for the non-stimulated M1. A higher ISP value indicates a higher inhibitory flow from the non-stimulated M1 to the stimulated M1.
Interhemispheric signal propagation (ISP) in TMS-evoked potential. | At 3-month
  ISP measured using concurrent TMS-evoked potential is set as another outcome for measuring the interhemispheric inhibitory flow between the bilateral M1s. TMS-evoked activity will be defined as the local mean field power (LMFP) of six channels surrounding the M1 (Left: C1, C3, C5, CP1, CP3, CP5; Right: C2, C4, C6, CP2, CP4, CP6) in a specific time frame. Because of the approximately 10 ms of transcallosal conduction, the LMFP from 50 to 130 ms is rectified for the stimulated M1 and from 60 to 140 ms for the non-stimulated M1. A higher ISP value indicates a higher inhibitory flow from the non-stimulated M1 to the stimulated M1.

IPD SHARING:
Plan to Share IPD: Undecided